CLINICAL TRIAL: NCT06561568
Title: Additional Effects of Kinesio Taping on Knee Joint Proprioception and Spatiotemporal Gait Parameters in Patient With Chrondromalacia Patellae
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/20
Record Dates: First submitted 2024-07-30; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Chondromalacia
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. KInesio taping along with conventional physical therapy will be applied in one group and the second will receive conventional physical therapy only. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy (exercise therapy) group (Active Comparator): Group A will receive this conventional physical therapy protocol for chondromalacia patellae
  * they will perform stretches to warm up and cool down. Resistance training ,in which patient will perform each exercise for 3 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
  * Frequency: 3 times a week for 4 weeks.
  Interventions: Diagnostic Test: Conventional physical therapy
- Kinesio taping + Conventional physical therapy group (Experimental): Group B will be given kinesio taping with conventional physical therapy protocol for chondromalacia patellae.
  .Kinesio tape will be applied on Vastus medialis Oblique and around the patella.
  • Frequency: 3 times a week for 4 weeks. They will perform stretches to warm up and cool down. Resistance training ,in which patient will perform each exercise for 3 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
  Frequency: 3 times a week for 4 weeks.
  Interventions: Diagnostic Test: Conventional physical therapy; Other: Kinesiotaping

INTERVENTIONS:
Diagnostic Test: Conventional physical therapy — Conventional physical therapy protocol for chondromalacia patellae consist of stretches to warm up and cool down Resistance training ,in which patient will perform each exercise for 3 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
Other: Kinesiotaping — Kinesio tape will be applied on Vastus medialis Oblique and around the patella.
  • Frequency: 3 times a week for 4 weeks.
  Arms: Kinesio taping + Conventional physical therapy group

SUMMARY:
Chondromalacia patellae (CMP), also known as runner's knee, is characterized by anterior knee pain (AKP) and typically occurs in youngsters. Causes of chondromalacia patellae include micro trauma wear and tear, post traumatic injuries and muscular imbalance. In Chondromalacia patella pain is behind or around the patella caused by stress in the patellofemoral joint that usually provoked by climbing stairs, squatting, and sitting with flexed knees for longer time periods. Patients of CMP presents with patellar mal-tracking, muscular weakness, proprioceptive deficit. Exercise training has been proven beneficial for CMP patients but additive effect of kinesio taping along with exercise have not been seen yet in these patients. The study will help people with chondromalacia patellae to improve their quality of life. The findings will contribute to future research in chondromalacia patellae management.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age: Under 60yrs
* Pain while stair climbing, kneeling, squatting, changing position from sitting to standing and running

Exclusive criteria:

* Instability of tibiofemoral joint
* Subluxation of patellofemoral joint
* Patellar instability
* Previous surgery of lower limb
* Positive findings on examination of knee ligaments, menisci and bursa.

Exclusion Criteria:

-

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proprioception | 4 weeks
  Proprioception will be measured using goniometer.
Pain intensity | 4 weeks
  Pain will be measured using numeric pain rating scale (NPRS) It is a self-rated scale where patient rate their pain from 0-10. 0 shows no pain where 10 shows worst pain.
Functional status | 4 weeks
  Functional status is assessed by lower extremity functional scale LEFS. The LEFS is scored on a scale of 0 to 80, with higher scores indicating better lower limb function. The interpretation of the scores is based on following categories. 0-20 Severe Functional limitation.21-40 moderate functional limitation and 41 and above is good functional status.
Gait Speed | 4 Weeks
  Gait analysis will be done to analyze speed.. A greater speed signifies positive outcome and prognosis. Speed = distance(m) x time(s)
Gait cadence | 4 Weeks
  Gait analysis will be done to analyze cadence. A greater cadence signifies positive outcome and prognosis. Cadence(steps/min) = steps countedx60/ time(s)
Gait cycle time | 4 weeks
  Gait analysis will be done to analyze cycle time. A greater cycle time signifies positive outcome and prognosis. Cycle time(s)=time(s) x2/steps counted
Stride length | 4 weeks
  Gait analysis will be done to analyze stride length. A greater stride length signifies positive outcome and prognosis. Stride Length(m)=Speed(m/s)xcycle time(s)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Pakistan